CLINICAL TRIAL: NCT00537771
Title: A Prospective, Randomized, Multicentre, Comparative and Open-label Study on Hepatotoxicity of ARIMIDEX Compared With Tamoxifen in Adjuvant Therapy in Postmenopausal Women With Hormone Receptor+ Early Breast Cancer
Brief Title: Liver Safety Under Upfront Arimidex vs Tamoxifen
Acronym: HEART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D5392L00023
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Early Breast cancer; adjuvant therapy; hormone receptor; hormonal therapy; anastrozole; tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Anastrozole (ARIMIDEX)
  Interventions: Drug: Anastrozole
- 2 (Active Comparator): Tamoxifen
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — 1 mg once daily oral dose
  Other Names: ARIMIDEX; ZD1033
  Arms: 1
Drug: Tamoxifen — 20 mg once daily oral dose
  Other Names: NOLVADEX
  Arms: 2

SUMMARY:
The primary objective is to compare ARIMIDEX (anastrozole) 1 mg once daily with Tamoxifen 20 mg once daily as adjuvant treatment in terms of: incidence of fatty liver diseases.

The second objectives are to compare ARIMIDEX (anastrozole) 1 mg once daily with Tamoxifen 20 mg once daily as adjuvant treatment in terms of: incidences of abnormal liver function test, and time to treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven HR+ invasive breast cancer
* Completed all primary surgery and chemotherapy (if given), and were candidates to receive hormonal adjuvant therapy
* Postmenopausal woman

Exclusion Criteria:

* clinical evidence of metastatic disease
* previous adjuvant hormonal therapy for breast cancer
* liver diseases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Gu, Study Director — AstraZeneca; Fengping Liang, Study Chair — AstraZeneca; Prof. Wang Shenming, Principal Investigator — AstraZeneca
Locations (16):
- China (16):
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Wuchang, Hubei
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Dalian, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xian, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Tianjin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in 28 centres in the People's Republic of China. FSI: 18Sep2007; LSI: 28 Feb2009;LSLV:20 Dec 2011.
Pre-assignment Details: A total of 384 patients were screened (informed consent signed and CRF started) and 353 patients were randomized with 175 patients in the Tamoxifen group and 178 in the Arimidex group.
Groups:
- Arimidex Group: Anastrozole(ARIMIDEX): 1 mg once daily oral dose
- TAM Group: Tamoxifen : 20 mg once daily oral dose
Period: Overall Study
Arm/Group | Arimidex Group | TAM Group
Started | 178 | 175
Completed | 149 | 114
Not Completed | 29 | 61
Not completed — Withdrawal by Subject | 6 | 23
Not completed — Adverse Event | 8 | 15
Not completed — Lost to Follow-up | 9 | 15
Not completed — Protocol Violation | 2 | 6
Not completed — Severe Non-Compliance to Protocol | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arimidex Group | TAM Group | Total
Number analyzed (Participants) | 178 | 175 | 353
Age Continuous [Mean (Standard Deviation); unit: years] | 59.7 (7.77) | 59.4 (8.84) | 59.6 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 175 | 353
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Fatty Liver Disease
Description: The primary objective is to compare ARIMIDEX (anastrozole) 1 mg once daily with Tamoxifen 20 mg once daily as adjuvant treatment in terms of: incidence of fatty liver diseases.
Time Frame: At 48 weeks, 96 weeks, 144 weeks
Measure: Number; unit: participants
Arm/Group | Arimidex Group | TAM Group
Number analyzed (Participants) | 178 | 175
participants
  48 weeks | 9 | 53
  96 weeks | 15 | 66
  144 weeks | 26 | 72

2. Secondary Outcome: Incidence of Abnormal Liver Function
Description: The second objectives are to compare ARIMIDEX (anastrozole) 1 mg once daily with Tamoxifen 20 mg once daily as adjuvant treatment in terms of: incidences of abnormal liver function test, and time to treatment failure.
Time Frame: At 48 weeks, 96 weeks, 144 weeks
Measure: Number; unit: participants
Arm/Group | Arimidex Group | TAM Group
Number analyzed (Participants) | 178 | 175
participants
  48 weeks | 29 | 36
  96 weeks | 37 | 40
  144 weeks | 44 | 43

3. Secondary Outcome: Time to Treatment Failure
Time Frame: Within 3 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arimidex Group | TAM Group
Number analyzed (Participants) | 178 | 175
days | 1112 [1053 to NA] — The upper limit of 95% Confidence Interval for Median of Time to treatment failure was substantially longer than 1122 and was not observed during the trial period. | 454 [353 to 673]

ADVERSE EVENTS:
Arm/Group | Arimidex Group | TAM Group
Serious Adverse Events (participants affected / at risk) | 4/178 | 4/175
Other Adverse Events (participants affected / at risk) | 39/178 | 41/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimidex Group (N=178) | TAM Group (N=175)
Fall (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Cervicitis (Infections and infestations) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Uterine atony (Reproductive system and breast disorders) | 0 | 1
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arimidex Group (N=178) | TAM Group (N=175)
Endometrial Hypertrophy (Reproductive system and breast disorders) | 0 | 10
Vaginal discharge (Reproductive system and breast disorders) | 1 | 9
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 4
Nasopharyngitis (Infections and infestations) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less